CLINICAL TRIAL: NCT01896414
Title: Metabolic Actions of Omega-3 Fatty Acids on Inflammation and Adipocyte Lipolysis in the Metabolic Syndrome
Brief Title: Metabolic Actions of Omega-3 Fatty Acids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institutes of Health (NIH) (NIH); US Department of Veterans Affairs (U.S. Federal Agency); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michael Miller, Cardiologist, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HP-00052080; R21HL113576-01 (NIH)
Record Dates: First submitted 2013-06-18; First posted 2013-07-11 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Omega 3 Fish Oil
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPA (marine fatty acids) (Experimental): Subjects will receive EPA , four 1 gram capsules daily.
  Interventions: Dietary Supplement: EPA (marine fatty acids)
- Placebo (Placebo Comparator): Subjects will be randomized to receive placebo, four 1 gram capsules daily.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: EPA (marine fatty acids) — Subjects will be randomized to receive either EPA or placebo, four 1 gram capsules daily.
  Arms: EPA (marine fatty acids)
Dietary Supplement: Placebo — Subjects will be randomized to receive either EPA/ or placebo, four 1 gram capsules daily.
  Arms: Placebo

SUMMARY:
The metabolic syndrome raises the risk of heart disease and is currently at epidemic proportions in the U.S. It consists of 3 of the following components: central obesity, high triglycerides, low HDL, abnormal blood pressure and impaired fasting glucose levels. Previous studies have suggested that omega-3 fish oil may influence some of these components but the mechanisms involved are not well understood. Therefore, this proposal will investigate how omega-3 fish oils affect inflammation, lipids and fat breakdown by comparing it to placebo. Favorable outcomes from this study could translate into a new approach to improve heart disease risk in men and women with the metabolic syndrome.

DETAILED DESCRIPTION:
Metabolic Actions of Omega-3 Fatty Acids on Inflammation and Adipocyte Lipolysis in the Metabolic Syndrome

Epidemiological studies identify metabolic syndrome (MetS) as a biomarker of cardiovascular disease (CVD) risk, and recent AHA scientific statements recommend intensive lifestyle diet and exercise measures to reduce risk. Marine-derived omega-3 polyunsaturated fatty acids such as, eicosapentanoic acid (EPA) improve many constituents of the metabolic syndrome such as lowering fasting TG and glucose levels, inflammation, insulin resistance and blood pressure. These improvements may be mediated by increased fat cell storage and metabolism and lipids, reducing inflammation and ectopic fat deposition in visceral abdominal tissue, muscle and liver that results in excessive pro-inflammatory intra-abdominal fat (IAF), insulin resistance and reduced levels of HDL cholesterol, hallmark characteristics of the MetS. The anti-inflammatory actions of EPA lower acute phase reactants (APRs) and proinflammatory mediators are mechanisms for their lipid lowering and insulin sensitizing effects to reduce CVD risk. The systematic investigation of marine-derived omega-3 PUFAs on these inflammatory, metabolic and physiological parameters will provide new mechanistic insights for the therapeutic use of a potentially beneficial, safe nutraceutical, EPA in patients with MetS. Thus, it is our hypothesis that supplementation of marine-derived omega-3 PUFAs, will reduce constituents of MetS as well as systemic and tissue inflammation, insulin resistance (HOMA-IR), adipocyte lipolysis and cytokine release from AT to enhance TG storage capacity of subcutaneous AT. The reduction in inflammation and increase in insulin sensitivity will remodel adipose tissue to function more efficiently in TG uptake and storage; thus, reducing circulating FFAs and cytokines. We postulate that these metabolic effects may decrease ectopic fat deposition in viscera (IAF and muscle), an intriguing, novel outcome that provides rationale for the 9 month treatment.

The Specific Aims are to conduct a pilot 9 month randomized trial in adults with high Tg and at least one other component of the MetS to compare the effects of EPA vs. placebo on:

Aim 1: Metabolic (e.g., lipoproteins, inflammatory cytokines, acute phase reactants, glucose tolerance/insulin resistance) and adipose tissue responses (basal and insulin suppression of lipolysis (ED50), LPL activity, cytokine release and lipogenesis).

Aim 2: Regional fat distribution quantified anthropometrically as waist and hip circumference, visceral and subcutaneous adipose volumes and muscle lipid accumulation by CT-scan and body composition (total and regional fat mass) by dual energy absorptiometry (DXA).

These outcomes have potentially intriguing therapeutic implications for marine derived omega-3 PUFA supplementation as part of a lifestyle program for patients at increased cardiometabolic risk.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic Syndrome, including 2 of the following:

  1. Treated Hyperlipidemia or Untreated Triglycerides > 150 mg/dL
  2. Waist circumference (inches) > 35 (women) or >40 (men)
* And at least 1 additional factor:
* Treated Hypertension or Untreated Blood pressure >130/85 and < 160/100 mm Hg
* HDL-C < 40 mg/dL men < 50 mg/dL women
* Glucose > 100mg/dL and HbA1c < 6.1%

Exclusion Criteria:

* Fasting TG > 500 mg/dL or LDL > 180 mg/dL
* Fasting glucose> 125 mg/dL or history of diabetes mellitus
* Hematologic or malignant disorders
* Morbid Obesity (BMI > 50 kg/m2)
* Endocrine (thyroid) or metabolic disorders (unless treated and under control)
* Alcohol consumption greater than (2) 4-ounce glasses of table wine, (2) 12-oz bottles of beer or 2 shots of spirits in men or women
* Active IV drug abuse within the past 6 months
* Clinical depression (per PI evaluation)
* Immunosuppressive or other therapy that would interfere with research testing

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07; Primary Completion 2016-05-30 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
Biochemical measurements of lipids, glucose homeostasis, inflammatory markers, and adipocyte responses to mediators of lipolysis | Up to 2 years
  Metabolic (e.g., lipoproteins, inflammatory cytokines, acute phase reactants, glucose tolerance/insulin resistance) and adipose tissue responses (basal and insulin suppression of lipolysis (ED50), LPL activity, cytokine release and lipogenesis).

SECONDARY OUTCOMES:
Determination of regional fat distribution, visceral and subcutaneous adipose volume and body composition | Up to 2 years
  Regional fat distribution quantified anthropometrically as waist and hip circumference, visceral and subcutaneous adipose volumes and muscle lipid accumulation by CT-scan and body composition (total and regional fat mass) by dual energy absorptiometry (DXA).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Miller, M.D., Principal Investigator — University of Maryland, College Park
Locations (2):
- United States (2):
  - University of Maryland Medical Center, Baltimore, Maryland
  - Amish Research Center, Lancaster, Pennsylvania